CLINICAL TRIAL: NCT01501617
Title: The Clinical Effects of HSC (Hair Stimulating Complex) on Hair Growth in Androgenetic Alopecia: A Phase I/II Clinical Trial
Brief Title: Safety and Efficacy of Hair Stimulating Complex (HSC) on Hair Growth in Males With Androgenetic Alopecia
Acronym: HSC Phase I/II
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Histogen (Industry)
Collaborators: Gleneagles CRC Pte Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-HIS006-PH
Record Dates: First submitted 2011-12-22; First posted 2011-12-29 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Androgenetic Alopecia
Keywords: Hair Loss; Androgenetic Alopecia; Baldness; Male pattern baldness; Male pattern hair loss; Hair Regrowth; Alopecia; Hair growth; Regrow Hair
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HSC- Hair Stimulating Complex (Experimental): Hair Stimulating Complex will be injected intradermally into the scalp of the test subject at 2 timepoints (Baseline and 6 Weeks after Baseline) using sterile syringes with 30 gauge needles at a volume of 0.1 mL per injection. A total of 8 injections (about 3mm apart) will be administered into one of the the 2 randomized sites (left or right) of the subject's scalp. Six weeks after the Baseline injection, the same treatment site will receive a repeat dose (the same volume and number of injections as used in the baseline) with no crossover.
  Interventions: Biological: Hair Stimulating Complex (HSC)
- Dulbecco's Modified Eagle Medium, DMEM (Placebo Comparator): Dulbecco's Modified Eagle Medium (DMEM) will be administered the same way as described above into treatment zone of the test subject's scalp not treated with HSC.
  Interventions: Device: Dulbecco's Modified Eagle Medium, DMEM

INTERVENTIONS:
Biological: Hair Stimulating Complex (HSC) — Study preparation (experimental) of 0.8 mL will be injected intradermally at Baseline and Week 6.
  Arms: HSC- Hair Stimulating Complex
Device: Dulbecco's Modified Eagle Medium, DMEM — Study preparation (placebo comparator) of 0.8 mL will be injected intradermally at Baseline and Week 6.
  Arms: Dulbecco's Modified Eagle Medium, DMEM

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy in relation to dosing in the administration of Hair Stimulating Complex (HSC) in healthy men. HSC will be injected intradermally in the scalps of men with male pattern baldness (i.e. androgenetic alopecia).

DETAILED DESCRIPTION:
HSC consists of proteins secreted by human dermal cells under proprietary culture conditions that include reduced oxygen and bioreactors. Under these conditions, the cells secrete soluble proteins that include both growth factors and soluble precursors to the deposited extracellular matrix. Several of these proteins are known to be important in the control of the hair cycle and will stimulate resting hair follicles to resume hair formation.

ELIGIBILITY:
Inclusion Criteria:

1. Male, ages 21-65 years.
2. A healthy scalp with no cutaneous disorder.
3. Subject should be in good general health.
4. Male subjects must be classified 3 Vertex, 4, 4A (if large enough), 5, 5A, or 6 under the Norwood-Hamilton Classification for Male Pattern Hair Loss (See Appendix 1).
5. Subject must be Fitzpatrick Type I, II, III and IV skin pigmentation (See Appendix 2). Type IV is acceptable however Type I-III is preferable.
6. Willing and able to comply with scheduled visits (Total: 7 visits in 48 weeks)
7. Willing to maintain the same hair style during the study period.
8. Willing to have a total of four microscopic dot tattoos. Two tattoos per treatment site (one in the center and one on the edge) of the two target regions of the scalp at miniaturization zone.
9. Willing to have 2 cm2 hairs clipped at treatment areas.
10. Willing to forgo the use of scalp products, including dye, throughout the study except for study related dye.
11. Willing to use a mild, a non-ionic shampoo throughout the course of the study.

Exclusion Criteria:

1. History of keloid formation or hyperpigmentation.
2. A history of any acute or chronic illness that in the opinion of the investigators might confound the results of the study including some drugs or medications.
3. Active skin diseases (e.g. eczema, atopic dermatitis, psoriasis, skin cancer, sun damaged skin with actinic keratosis on scalp, etc.).
4. Routine high dosage use of anti-inflammatory medications (aspirin, ibuprofen, corticosteroids), immunosuppressive drugs or antihistamine medications (steroid nose drops and/or eye drops are permitted). Two 81 mg or one 325 mg aspirin per day is also acceptable.
5. Use of topical drugs or other cosmetics on the scalp.
6. Immunological disorders such as HIV positive, alopecia areata, and systemic lupus erythematosus.
7. Participation in any clinical study within the last four weeks.
8. Moderate or severe seborrheic dermatitis of scalp.
9. Damaged skin in or around test sites including sunburn, uneven skin tones, tattoos, scars or other disfiguration of the test site.
10. Use of OTC (over-the-counter) or prescriptive topical or hair treatments, as well as hair transplantation surgery during the last 6 months. This includes Minoxidil 2% or 5% and/or Finasteride 1mg or any 5alpha-reductase inhibitors.
11. Currently using hair system or wig.
12. Presence of hair transplants or scalp surgery.
13. History of allergy or intolerance to lidocaine and/or epinephrine.
14. Use of hair dye (not study related) during the study duration.
15. Any condition for which the Investigator determines that the subject could be placed under undue risk.
16. Reported history of allergy or intolerance to bovine proteins.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Systemic safety measures will be assessed by measuring vital signs, adverse experiences, laboratory tests (hematology, clinical chemistry and urinalysis)and immunological response (anti-drug antibodies) | Clinically significant change from screening visit to Week 12
Non-vellus hair counts | Change from Baseline to week 12 in treatment areas

SECONDARY OUTCOMES:
Hair Thickness Density | Change from Baseline to week 48 in treatment areas
Local safety measures will be assessed by clinical exam of treatment areas and monitoring adverse events | Clinically significant change from Screening visit to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Marie Reyes-Cacas, MD, Principal Investigator — The Medical City; Julieta P. Arambulo, MD, Principal Investigator — The Medical City
Locations (1):
- The Medical City, Pasig, Manila, Philippines